CLINICAL TRIAL: NCT01838122
Title: Prevalence of HbA1C in Different Categories of Obesity in Women With PCOS'A Propective Randomized Control Study
Brief Title: Prevalence of HbA1C in Women With PCOS
Acronym: WHI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Southern Cross Fertility Centre (Other)
Responsible Party: Principal Investigator, M.R. Bharucha, Faram E.Irani, Southern Cross Fertility Centre
Other Study IDs: HbA1C-PCOS; PCOS-IR (Registry Identifier: ICMJE)
Record Dates: First submitted 2013-04-15; First posted 2013-04-23 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Polycystic Ovarian Syndrome; Pelvic Endometriosis; Insulin Resistance; Non-insulin Dependent Diabetes Mellitus; Tubal Obstruction
Keywords: PCOS; HbA1C; Insulin resistance; OGTT; HOMA-IR; HOMA-B-cell
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Diabetes Mellitus, Type 2; Fallopian Tube Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Study Arm: This group/cohort will have subjects having infertility due to PCOS (as per Rotterdam criteria)
- Control arm: This group/cohort will have subjects without PCOS but with any other diagnosis of infertility or any other complain.

SUMMARY:
Women with PCOS have been observed to be potential diabetics.Recently,American Diabetes Association has suggested screening of women with PCOS for HbA1C.

DETAILED DESCRIPTION:
In view of recent suggestion of American Diabetes Association(ADA)to screen women with PCOS for HbA1C,we intend to study its prevalence in all categories of obesity in women with PCOS.

Women with PCOS by Rotterdam criteria will be screened for insulin resistance by using different techniques or tests.

Further, the sensitivity and specificity of HbA1C will be compared with sensitivity and specificity of other insulin resistance markers such as OGTT, Free androgen index, free testosterone, fasting insulin to glucose ratio, HOMA-IR and HOMA-B-CELL.

ELIGIBILITY:
Inclusion Criteria:

1. BMI of 25-35 Kg/Mt2
2. Atleast three of the Rotterdam criteria for diagnosis of PCOS.
3. Subjects with well stabilized Thyroid,if they had documented evidence of previousthyroid disorder.

Exclusion Criteria:

1. Subjects with documented diagnosis of Metabolic Syndrome.
2. Subjects with laparocopic and histopathologic diagnosis of Endometriosis. 3Subjects with Primary hyperprolectineamia.

4.Subjects with basal FSH >/=15mIU/ml. 5.Subjects with continuously elevated 17-0h-p.

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This population will have subjects with diagnosis of PCOS,by Rotterdam criteria regardless of complain(s)
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-09 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence of HbA1C in both arms of the cohort of subjects | September 2013
  HbA1C has been suggested as a potential marker for NIDDM in subjects with PCOS

CONTACTS AND LOCATIONS:
Overall Officials: Manchi R Bharucha, Ph.D, Study Director — Southern Cross Fertility Centre; Manchi R Bharucha, Ph.D., Study Director — Souther Cross Fertility Centre
Locations (1):
- Southern Cross Fertility Centre, Mumbai, Maharashtra, India

REFERENCES:
- [Result] Kim JJ, Choi YM, Cho YM, Jung HS, Chae SJ, Hwang KR, Hwang SS, Ku SY, Kim SH, Kim JG, Moon SY. Prevalence of elevated glycated hemoglobin in women with polycystic ovary syndrome. Hum Reprod. 2012 May;27(5):1439-44. doi: 10.1093/humrep/des039. Epub 2012 Feb 21. PMID 22357766